CLINICAL TRIAL: NCT03243656
Title: Randomized Clinical Trial of the Use of & Cyclosporine in Children With Sever Idiopathic Aplastic Anemia
Brief Title: Eltrombopag & Cyclosporine in Children With Sever Aplastic Anemia
Acronym: Eltroplastic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Ali Abdelfatah Ahmed, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAAhmed
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Eltrombopag
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- historical group (No Intervention): Immunosuppressive therapy (cyclosporine alone ),
- case arm (Active Comparator): cyclosporine plus an oral dose of Eltrombopag
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — An oral thrombopoietin receptor agonist
  Other Names: Revolade
  Arms: case arm

SUMMARY:
Aplastic anemia is a rare disorder characterized by pancytopenia and a hypo cellular bone marrow.but,It is very serious disease causing morbidity and mortality.

Aplastic anemia can be treated effectively with haematopoietic stem cell transplantation and immunosuppressive drug regimens but haematopoietic stem cell transplantation has limitations due to its cost and many patient are unsuitable. Immunosuppressive drug has a significant number of patients have persistent cytopenias. Currently, the treatment of these patients is regular transfusion, which are expensive, inconvenient, and associated with serious side effects related to iron overload and transfusion.

Eltrombopag is an oral thrombopoietin mimetic that selectively binds at the transmembrane and juxtamembrane domains of the thrombopoietin receptor, at sites distinct from the binding site of thrombopoietin therefore it does not compete for binding with the native molecule. It promoting thrombopoiesis and release of platelets from mature megakaryocytes. Also, promote other hematopoietic stem cell as well as in thrombopoiesis .

DETAILED DESCRIPTION:
Aplastic anemia is a rare disorder characterized by pancytopenia and a hypo cellular bone marrow.This causes a deficiency of all three blood cell types (pancytopenia): red blood cells (anemia), white blood cells (leukopenia), and platelets (thrombocytopenia) . The clinical consequences are anemia, usually with a requirement for frequent red blood cell transfusions, life-threatening bleeding from thrombocytopenia, and infection because of neutropenia. Bacterial and fungal infections are most common and are a significant cause of morbidity and mortality.

The incidence of acquired Aplastic anemia in Europe and North America is around two per million children per year . The incidence is 2-3 times higher in East Asia. There is no significant difference in incidence between males and females .

The pathogenesis of Aplastic anemia is complex and involves an abnormal hematopoietic microenvironment, hematopoietic stem cell/progenitor cell deficiencies and immunity disorders. The etiological basis for marrow failure includes primary defects in or damage to the stem cell or the marrow microenvironment. The distinction between acquired and inherited disease may present a clinical challenge, Congenital or inherited causes of Aplastic anemia are responsible for at least 25% of children with this condition and for perhaps up to 10% of adults. Acquired causes of Aplastic anemia form (80%) of cases, include Idiopathic (> 80 %), Post-infectious 15% (particularly after hepatitis 9%, Epstein-Barr virus , human immune deficiency virus, parvovirus, and mycobacteria, Drug-induced and toxins (4%).

Definitive and potentially curative therapy with haematopoietic stem cell transplantation However, only a minority (30 %) of patients have a suitable donor. Immunosuppressive therapy with horse or rabbit antithymocyte globulin plus cyclosporine is the most commonly used alternative treatment in about two thirds of cases. Response is associated with a favorable long-term outlook. 30 -40% of patients are refractory to immunosuppressive therapy and remain pancytopenic after therapy. Even patients that respond to immunosuppressive therapies with an improvement in their life-threatening neutropenia sometimes have persistent thrombocytopenia .

Aplastic anemia can be treated effectively with haematopoietic stem cell transplantation and immunosuppressive drug regimens but haematopoietic stem cell transplantation has limitations due to its cost and many patient are unsuitable. Immunosuppressive drug has a significant number of patients have persistent cytopenias. Currently, the treatment of these patients is regular transfusion, which are expensive, inconvenient, and associated with serious side effects related to iron overload and transfusion.

Thrombopoietin is a glycoprotein class 1 hematopoietic cytokine, produced primarily in the liver. It is a critical regulator of hematopoiesis. It acts through the thrombopoietin receptor which is expressed on hematopoietic stem and progenitor cells. Action results in a number of signal transduction events that prevent apoptosis, improve cell viability, promote growth, and possibly increase differentiation.

Eltrombopag is an oral thrombopoietin mimetic that selectively binds at the transmembrane and juxtamembrane domains of the thrombopoietin receptor, at sites distinct from the binding site of thrombopoietin therefore it does not compete for binding with the native molecule. It promoting thrombopoiesis and release of platelets from mature megakaryocytes. Also, promote other hematopoietic stem cell as well as in thrombopoiesis .Eltrombopag became the first oral platelet growth factor to receive Food and Drug Administration approval in 2008. This initial indication was for adult patients with chronic immune thrombocytopenic purpura. In 24 August 2015, this indication was extended to children age 1 to 17 with the same condition. In addition, it has been recently shown to be efficacious in the setting of aplastic anemia with trilineage responses in some patients and many achieving transfusion independence. It has license by the European Medicines Agency for this indication in August 2015. In 2017, the National Institutes of Health made Eltrombopag a standard of care in Aplastic anemia

ELIGIBILITY:
Inclusion Criteria:

Current diagnosis of sever Aplastic anemia

* Diagnosis of sever Aplastic anemia is established if Bone marrow cellularity <25% or and at least two of the following criteria are met:- (i) absolute neutrophil count less than 0.5 × 109/L, (ii) platelet count less than 20 × 109/L, and (iii) reticulocyte count less than 20 × 109/L
* No, evidence of viral or drug suppression of the marrow, dysplasia, or underproduction anemias secondary to B12, folate, iron or other reversible causes.
* Age equal to 1 years old to 18 years old
* Written informed consent signed by a parent or legal guardian prior to initiation of any study specific procedure.
* Hematopoietic stem cell transplantation is not available or suitable as a treatment option or has been refused by the patient.
* Bone marrow aspirate and biopsy at any time during the 4 weeks prior to first dose of eltrombopag

Exclusion Criteria:

Prior and/or active medical history of:-

* Fanconi anemia (via chromosomal breakage test or growth arrest by flow cytometry). Other known underlying congenital/inherited marrow failure syndromes.
* Symptomatic Paroxysmal Nocturnal Hemoglobinuria
* Other known or suspected underlying primary immunodeficiency
* Any malignancy
* Active infection not responding to appropriate therapy
* Any out of range lab values Creatinine >2.5 mg/dL× the upper limit of normal, Total bilirubin >1.5 × the upper limit of normal mg/dL ,Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 × the upper limit of normal
* Hypersensitivity to eltrombopag or its components
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
changes in Platelet count (at Baseline, 26 Weeks and up to 52 week) | 52 week
  increase of platelet count from baseline by 20,000/microliter or more (in the absence of platelet transfusion), or independence from platelet transfusions for a minimum of 8 weeks in patients who were previously transfusion-dependent.
Changes in hemoglobin count (at Baseline, 26 Weeks and up to 52 week) | 52 week
  measuring the following: Increase from baseline by 1.5 gram g/dL or more when the baseline hemoglobin level is <8.5 g/dL and no red blood cell (RBC) transfusion at baseline. A decrease of at least four units in RBC transfusions in the post-treatment 8-week period compared to the pre-treatment 8-week period..
changes in absolute Neutrophil count (at Baseline, 26 Weeks and up to 52 week) | 52 week
  measuring the increase in the absolute neutrophil count of more than 500 per cubic millimeter
complete response (CR) - 12 month | 52 weeks
  CR defined as all three parameters meet the following criteria : Hb ≥100 g/l, platelet count ≥100 × 109/L, and ANC ≥1 × 109/L. Additionally, patients had to be transfusion and growth factor independent
Partial response (PR) - 12 month | 52 weeks
  PR was defined as blood count no longer meeting Camitta criteria for severs aplastic anemia in case of sever aplastic anemia (SAA): Absolute neutrophil count (ANC) >500/μL Platelet count >20 000/μL Reticulocyte count >20 000/μL

SECONDARY OUTCOMES:
The hematological responses | up to to 52 week
  Duration of hematologic response Time from the date of the start of response to the date of relapse defined as again meeting criteria for severe or moderate aplastic anemia Duration of platelet and blood transfusion independence Transfusion independency is defined when blood and platelet transfusions are not required in a consecutive 8-week period. Transfusion dependency will be defined as at least 2 units of red blood cells or five units of random platelets or equivalent apheresis per month for a period of 8 weeks. The duration of platelet and blood transfusion independence will be evaluated separately.
The toxicity | Up to 30 days after last dose of study treatment
  Number of participants with adverse events Measure toxicity, using CTCAE associated with assessment of eltrombopag use, dose, and tolerability in patients with sever to very severe aplastic anemia
complete response (CR)- 6 month | 26 week
  CR defined as all three parameters meet the following criteria : Hb ≥100 g/l, platelet count ≥100 × 109/L, and ANC ≥1 × 109/L. Additionally, patients had to be transfusion and growth factor independent
Partial response (PR) - 6 month | 26 week
  PR was defined as blood count no longer meeting Camitta criteria for severs aplastic anemia in case of SAA.
  Absolute neutrophil count (ANC) >500/μL Platelet count >20 000/μL Reticulocyte count >20 000/μL
Overall hematologic response (CR + PR) rate - 6 month | 26 week
  Overall hematologic response = patients with complete response + patients with partial response .
  Partial response is defined as blood count no longer meeting Camitta criteria for severs aplastic anemia in case of SAA
  ANC >500/μL Platelet count >20 000/μL Reticulocyte count >20 000/μL
  Complete response is defined as all three parameters meet the following criteria:
  ANC > 1 000/μL Platelet count >100 000/μL Hemoglobin >10 g/L
Overall hematologic response (CR + PR) rate - 12 month | 52 week
  Overall hematologic response = patients with complete response + patients with partial response.
  Partial response is defined as blood count no longer meeting Camitta criteria for severs aplastic anemia in case of SAA
  ANC >500/μL Platelet count >20 000/μL Reticulocyte count >20 000/μL
  Complete response is defined as all three parameters meet the following criteria:
  ANC > 1 000/μL Platelet count >100 000/μL Hemoglobin >10 g/L

CONTACTS AND LOCATIONS:
Locations (1):
- Facility of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guinan EC. Acquired aplastic anemia in childhood. Hematol Oncol Clin North Am. 2009 Apr;23(2):171-91. doi: 10.1016/j.hoc.2009.01.011. PMID 19327578
- [Background] Young NS, Bacigalupo A, Marsh JC. Aplastic anemia: pathophysiology and treatment. Biol Blood Marrow Transplant. 2010 Jan;16(1 Suppl):S119-25. doi: 10.1016/j.bbmt.2009.09.013. Epub 2009 Sep 24. PMID 19782144
- [Background] Issaragrisil S, Kaufman DW, Anderson T, Chansung K, Leaverton PE, Shapiro S, Young NS. The epidemiology of aplastic anemia in Thailand. Blood. 2006 Feb 15;107(4):1299-307. doi: 10.1182/blood-2005-01-0161. Epub 2005 Oct 27. PMID 16254144
- [Background] Marsh JC, Mufti GJ. Eltrombopag: a stem cell cookie? Blood. 2014 Mar 20;123(12):1774-5. doi: 10.1182/blood-2014-02-553404. No abstract available. PMID 24652959
- [Background] Garnock-Jones KP, Keam SJ. Eltrombopag. Drugs. 2009;69(5):567-76. doi: 10.2165/00003495-200969050-00005. PMID 19368418
- [Background] Montane E, Ibanez L, Vidal X, Ballarin E, Puig R, Garcia N, Laporte JR; Catalan Group for Study of Agranulocytosis and Aplastic Anemia. Epidemiology of aplastic anemia: a prospective multicenter study. Haematologica. 2008 Apr;93(4):518-23. doi: 10.3324/haematol.12020. Epub 2008 Mar 5. PMID 18322256
- [Background] Qian H, Buza-Vidas N, Hyland CD, Jensen CT, Antonchuk J, Mansson R, Thoren LA, Ekblom M, Alexander WS, Jacobsen SE. Critical role of thrombopoietin in maintaining adult quiescent hematopoietic stem cells. Cell Stem Cell. 2007 Dec 13;1(6):671-84. doi: 10.1016/j.stem.2007.10.008. Epub 2007 Nov 20. PMID 18371408
- [Background] Kaushansky K. Historical review: megakaryopoiesis and thrombopoiesis. Blood. 2008 Feb 1;111(3):981-6. doi: 10.1182/blood-2007-05-088500. PMID 18223171
- [Background] Bussel JB, Cheng G, Saleh MN, Psaila B, Kovaleva L, Meddeb B, Kloczko J, Hassani H, Mayer B, Stone NL, Arning M, Provan D, Jenkins JM. Eltrombopag for the treatment of chronic idiopathic thrombocytopenic purpura. N Engl J Med. 2007 Nov 29;357(22):2237-47. doi: 10.1056/NEJMoa073275. PMID 18046028
- [Background] de Laval B, Pawlikowska P, Petit-Cocault L, Bilhou-Nabera C, Aubin-Houzelstein G, Souyri M, Pouzoulet F, Gaudry M, Porteu F. Thrombopoietin-increased DNA-PK-dependent DNA repair limits hematopoietic stem and progenitor cell mutagenesis in response to DNA damage. Cell Stem Cell. 2013 Jan 3;12(1):37-48. doi: 10.1016/j.stem.2012.10.012. Epub 2012 Dec 13. PMID 23246483
- [Background] Olnes MJ, Scheinberg P, Calvo KR, Desmond R, Tang Y, Dumitriu B, Parikh AR, Soto S, Biancotto A, Feng X, Lozier J, Wu CO, Young NS, Dunbar CE. Eltrombopag and improved hematopoiesis in refractory aplastic anemia. N Engl J Med. 2012 Jul 5;367(1):11-9. doi: 10.1056/NEJMoa1200931. PMID 22762314
- [Background] Desmond R, Townsley DM, Dumitriu B, Olnes MJ, Scheinberg P, Bevans M, Parikh AR, Broder K, Calvo KR, Wu CO, Young NS, Dunbar CE. Eltrombopag restores trilineage hematopoiesis in refractory severe aplastic anemia that can be sustained on discontinuation of drug. Blood. 2014 Mar 20;123(12):1818-25. doi: 10.1182/blood-2013-10-534743. Epub 2013 Dec 17. PMID 24345753
- [Background] Alter BP. Aplastic Anemia, Pediatric Aspects. Oncologist. 1996;1(6):361-366. PMID 10388017
- [Background] Ballmaier M, Germeshausen M, Krukemeier S, Welte K. Thrombopoietin is essential for the maintenance of normal hematopoiesis in humans: development of aplastic anemia in patients with congenital amegakaryocytic thrombocytopenia. Ann N Y Acad Sci. 2003 May;996:17-25. doi: 10.1111/j.1749-6632.2003.tb03228.x. PMID 12799278
- [Background] Dezern AE, Brodsky RA. Clinical management of aplastic anemia. Expert Rev Hematol. 2011 Apr;4(2):221-30. doi: 10.1586/ehm.11.11. PMID 21495931
- [Background] Gupta V, Eapen M, Brazauskas R, Carreras J, Aljurf M, Gale RP, Hale GA, Ilhan O, Passweg JR, Ringden O, Sabloff M, Schrezenmeier H, Socie G, Marsh JC. Impact of age on outcomes after bone marrow transplantation for acquired aplastic anemia using HLA-matched sibling donors. Haematologica. 2010 Dec;95(12):2119-25. doi: 10.3324/haematol.2010.026682. Epub 2010 Sep 17. PMID 20851870
- [Background] Marsh JC, Ball SE, Cavenagh J, Darbyshire P, Dokal I, Gordon-Smith EC, Keidan J, Laurie A, Martin A, Mercieca J, Killick SB, Stewart R, Yin JA; British Committee for Standards in Haematology. Guidelines for the diagnosis and management of aplastic anaemia. Br J Haematol. 2009 Oct;147(1):43-70. doi: 10.1111/j.1365-2141.2009.07842.x. Epub 2009 Aug 10. No abstract available. PMID 19673883
- [Background] Rauff B, Idrees M, Shah SA, Butt S, Butt AM, Ali L, Hussain A, Irshad-Ur-Rehman, Ali M. Hepatitis associated aplastic anemia: a review. Virol J. 2011 Feb 28;8:87. doi: 10.1186/1743-422X-8-87. PMID 21352606
- [Background] Young NS. Pathophysiologic mechanisms in acquired aplastic anemia. Hematology Am Soc Hematol Educ Program. 2006:72-7. doi: 10.1182/asheducation-2006.1.72. PMID 17124043
- [Background] Zhang J, Yang T. [Meta-analysis of association between organophosphorus pesticides and aplastic anemia]. Zhonghua Liu Xing Bing Xue Za Zhi. 2015 Sep;36(9):1005-9. Chinese. PMID 26814872
- [Background] Wu Y, Yu J, Zhang L, Luo Q, Xiao JW, Liu XM, Xian Y, Dai BT, Xu YH, Su YC. [Hematopoiesis support of mesenchymal stem cells in children with aplastic anemia]. Zhongguo Dang Dai Er Ke Za Zhi. 2008 Aug;10(4):455-9. Chinese. PMID 18706160
- [Background] Scheinberg P. Aplastic anemia: therapeutic updates in immunosuppression and transplantation. Hematology Am Soc Hematol Educ Program. 2012;2012:292-300. doi: 10.1182/asheducation-2012.1.292. PMID 23233595
- [Background] Scheinberg P, Nunez O, Weinstein B, Scheinberg P, Biancotto A, Wu CO, Young NS. Horse versus rabbit antithymocyte globulin in acquired aplastic anemia. N Engl J Med. 2011 Aug 4;365(5):430-8. doi: 10.1056/NEJMoa1103975. PMID 21812672
- [Background] Townsley DM, Scheinberg P, Winkler T, Desmond R, Dumitriu B, Rios O, Weinstein B, Valdez J, Lotter J, Feng X, Desierto M, Leuva H, Bevans M, Wu C, Larochelle A, Calvo KR, Dunbar CE, Young NS. Eltrombopag Added to Standard Immunosuppression for Aplastic Anemia. N Engl J Med. 2017 Apr 20;376(16):1540-1550. doi: 10.1056/NEJMoa1613878. PMID 28423296